CLINICAL TRIAL: NCT07347665
Title: Randomized Clinical Trial of Endovascular Therapy for Acute Ischemic Stroke With Occlusion of the M2 Segment of Middle Cerebral Artery (the Recovery by Endovascular Salvage for Cerebral Ultra-acute Embolism-M2 Occlusion Trial: RESCUE-M2O Trial)
Brief Title: Randomized Clinical Trial of Endovascular Therapy for Acute Ischemic Stroke With Occlusion of the M2 Segment of Middle Cerebral Artery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hyogo Medical University (Other)
Responsible Party: Principal Investigator, Kazutaka Uchida, Associate Professor (Stroke Center), Hyogo Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R000066936
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Endovascular Therapy; Acute Ischemic Stroke; Acute Ischemic Stroke (AIS) Related to a Distal Occlusion
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical therapy with endovascular therapy (Experimental)
  Interventions: Procedure: Endovascular therapy
- Medical therapy alone (No Intervention)

INTERVENTIONS:
Procedure: Endovascular therapy — Endovascular therapy for acute ischemic stroke with occlusion of the M2 segment of the middle cerebral artery.
  Arms: Medical therapy with endovascular therapy

SUMMARY:
RESCUE-M2O trial is a prospective, open label, blinded endpoint (PROBE), two-arm, randomized, controlled, post-market study to assess the efficacy and safety of endovascular therapy for acute ischemic stroke with occlusion of the M2 segment of the middle cerebral artery.

ELIGIBILITY:
Inclusion Criteria:

1. Acute cerebral infarction
2. Aged 18-84 years
3. NIHSS score at admission ≥ 8
4. Prestroke mRS scores of 0-1 (able to carry out all usual activities)
5. Occlusion of the M2 segment of MCA on digital subtraction angiography
6. ASPECTS ≥ 8 or DWI-ASPECTS ≥ 8
7. Ineligible or failed intravenous tPA (no recanalization within 30 min after injection)
8. Randomization can be completed within 24 h from the last known well time
9. EVT can be initiated within 30 min from randomization.
10. The patient or their legally authorized representative has signed the informed consent form.

Exclusion Criteria:

1. Occlusion of the anterior temporal artery, duplicate M1, or accessory M1
2. Occlusion of multiple major intracranial arteries
3. Difficulty in endovascular access due to tortuous vascular anatomy
4. Significant mass effect with midline shift on CT (or MRI)
5. Known allergy (more severe than skin rash) to contrast agents
6. Evidence of acute intracranial hemorrhage on CT (or MRI)
7. Pregnant or potentially pregnant
8. Clinical evidence of chronic occlusion
9. High risk of hemorrhage (platelet < 40,000/ul, APTT > 50 sec or PT-INR > 3.0)
10. Participating in any other therapeutic investigational trial
11. Judgment of the investigator to be non-compliant or uncooperative during the study

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Achievement of mRS scores of 0-2 | 90 days after randomization

SECONDARY OUTCOMES:
Achievement of mRS scores of 0-1 | 90 days after randomization
mRS shift analysis | 90 days after randomization
NIHSS improvement of 8 points or more | 48 hours after randomization
QOL (EQ-5D-3L) | 90 days after randomization
Symptomatic intracranial hemorrhage | 48 hours after randomization
Any intracranial hemorrhage | 48 hours after randomization
All cause death | 90 days after randomization
Recurrence of cerebral infarction | 90 days after randomization
Decompressive craniectomy | 7 days after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Hyogo Medical University, Nishinomiya, Hyōgo, Japan